CLINICAL TRIAL: NCT03813771
Title: Targeted Treatment Early With Etanercept Plus Methotrexate Versus T2T Care for DMARD-naïve Early RA Patients. A Prospective, Longitudinal Cohort Study With Embedded Pilot Randomised Controlled Trial to Assess Treatment Rationalisation Based on naïve T-cell Stratification.
Brief Title: Targeted Treatment Early With Etanercept + Methotrexate vs.T2T Care for DMARD-naïve Early RA Patients Based on naïve T-cell Stratification
Acronym: TEEMS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Leeds (Other)
Collaborators: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RR16/209; 2016-002344-16 (EudraCT Number)
Record Dates: First submitted 2018-09-12; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
Keywords: T-cells; Treat to Target; DMARD-naive; Benepali
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Sulfasalazine; Methotrexate; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal cohort study with an embedded pilot randomised controlled trial. Patients with normal naive T-cell status will receive standard T2T care with methotrexate. Patients with abnormal naive T-cell status will be randomised 1:1 to T2T care vs. Benepali + T2T care with methotrexate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Abnormal T-cells: Benepali + T2T Care (Experimental): Treatment Arm C will receive Benepali and methotrexate combination therapy and followed as per T2T care over a total duration of 24 weeks. Sulfasalazine or Hydroxychloroquine may be added to therapy at follow up visits in-line with T2T care.
  Benepali will be administered subcutaneously at a dose of 50mg weekly and discontinued at the primary endpoint (24 weeks).
  Methotrexate will be administered orally at a starting dose of 15mg weekly. It may be increased in line with T2T care (to a maximum of 25mg) over the 24 weeks.
  Interventions: Drug: Benepali; Drug: Methotrexate
- Abnormal T-cells: Methotrexate + T2T Care (Active Comparator): Treatment Arm B will receive initial methotrexate monotherapy with adoption of a treat to target protocol (standard care involving monthly DAS28-ESR assessment with escalation to combination synthetic DMARD (Including sulfasalazine and/or hydroxychloroquine).
  therapy if not achieving low disease activity (LDA) at, or after, 8 weeks).
  Interventions: Drug: Sulfasalazine; Drug: Methotrexate; Drug: Hydroxychloroquine
- Normal T-cells: Methotrexate + T2T Care (Other): Treatment Arm A will receive standard T2T care as per Arm B.
  Interventions: Drug: Sulfasalazine; Drug: Methotrexate; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Benepali — Benepali will be adminstered subcutaneously at a dose of 50mg weekly and discontinued at the primary endpoint (24 weeks).
  Other Names: Etanercept
  Arms: Abnormal T-cells: Benepali + T2T Care
Drug: Sulfasalazine — Sulfasalazine will be added at follow up visits (T2T care) if the subject fails to achieve low disease activity,administered orally at a dose of 1g twice daily.
  Arms: Abnormal T-cells: Methotrexate + T2T Care; Normal T-cells: Methotrexate + T2T Care
Drug: Methotrexate — Methotrexate will be administered orally at a starting dose of 15mg weekly. It may be increased in line with T2T care (to a maximum of 25mg) over the 24 weeks.
Drug: Hydroxychloroquine — Hydroxychloroquine will be added at follow up visits (T2T care) if the subject fails to achieve low diseaseactivity, administered at a dose of 200mg daily.
  Arms: Abnormal T-cells: Methotrexate + T2T Care; Normal T-cells: Methotrexate + T2T Care

SUMMARY:
The main aim of the study is to determine the clinical utility of naive T-cell stratification for rationalising treatment with methotrexate (MTX), for DMARD-naive early RA patients. Thus, it aims to determine whether TNFi therapy (Benepali) instituted as first-line therapy in DMARD-naive early RA patients with poor T-cell prognostication confers better outcomes (clinical, structural and immunological). Hence, this would enable early targeted treatment for those with a poorer prognosis based on their immunological status.

DETAILED DESCRIPTION:
The current optimal therapeutic approach in early RA is to start MTX to target inflammation and induce remission.Prediction of MTX therapy response remains a key clinical need to enable the identification of patients who would benefit from an alternative, more aggressive treatment strategy. Multiple predictors of remission with MTX have been reported over the years but none have entered routine clinical practice.

We previously reported that T-cell phenotyping at baseline could predict remission in DMARD-naïve early RA treated with MTX. Reduced naïve CD4+ T-cell frequency was the most predictive factor, using both a pilot and a replication cohort.These data confirmed the potential value of using naïve CD4+ T-cells as a biomarker of MTX induced remission in early RA.

The clinical utility of measuring T-cell subsets is therefore strongly indicated by these data and suggests that measurement of T- cell subsets can be used to rationalise the use of MTX as first-line therapy.Predicting response to MTX has important clinical value to identify patients who will do well on MTX but furthermore for directing those who will have a sub-optimal response to MTX to receive alternative therapy without any harmful delay and in line with the treat to target principle.

The current study aims to confirm/validate the clinical value of T-cell subset quantification for the prediction of MTX response in early RA, by stratified interventions based on baseline naïve CD4+ T-cell status.

This is a Single centre, phase IV, open-label, prospective, longitudinal cohort study with an embedded pilot randomised controlled trial that aims to assess whether MTX can be rationalised as a first-line treatment for DMARD-naïve early RA patients, according to baseline naïve CD4+ T-cell stratification.

Patients with newly diagnosed RA satisfying the inclusion criteria will be recruited from our early arthritis clinic. Eligible patients will be provided with written information on the study and will be given a minimum of 24 hours to read this information prior to being contacted by a research nurse (within one week). If interested they will be invited to a screening appointment within four weeks to confirm eligibility, obtain written consent and to collect the necessary clinical and laboratory data as per the study schedule. Following the screening visit, patients will attend a baseline assessment within four weeks.

Patients will be stratified based on their naïve CD4+ T-cell frequency (normal or abnormal based on our pre-defined cut-off values according to age and sex-matched controls). Patients with a normal T-cell frequency (Arm A) will commence MTX 15mg/week PO (+HCQ 400mg od) as per standard T2T practice. Follow-up (4, 12 and 24 weeks), dose escalation of MTX and treatment of flare will also be conducted in line with T2T care.

Patients with an abnormal T-cell frequency will be randomized 1:1 into 2 groups using randomly permuted block sizes and also followed up as per T2T care:

The first group (Arm B) will receive MTX 15mg/week PO (+HCQ 400mg od) The second group (Arm C) will receive MTX 15mg/week PO (+HCQ 400mg od) in combination with 50 mg subcutaneous Benepali® administered weekly.

Patients will be followed up for a period of 24 weeks and will undergo clinical, immunological and imaging assessments as stated in the study schedule. Following completion of the study, patients will either be followed up in our established inflammatory arthritis or biologics clinic. Patients in group C will discontinue their Benepali®.

This study will take place at the rheumatology out-patient department in Chapel Allerton Hospital, Leeds.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of RA as defined by the new ACR/EULAR 2010 classification criteria
* Newly diagnosed (within 12 weeks)
* Active disease at screening (DAS28ESR ≥3.2 or clinical evidence of synovitis)
* Anti-citrillunated protein antibody (ACPA) positive
* Male & female subjects ≥18 years old
* DMARD (disease modifying anti-rheumatic drug) naïve
* No use of intra-muscular, intra-articular or oral corticosteroids 4 weeks days prior to screening
* All male and female subjects biologically capable of having children must agree to use a reliable method of contraception for the duration of the study and 24 weeks after the end of the study period. Acceptable methods of contraception are surgical sterilisation, oral, implantable or injectable hormonal methods, intrauterine devices or barrier contraceptives.
* Patients must have the capacity and be willing to provide written informed consent and comply with the requirements of the protocol
* Subjects should be deemed to be in good health with respect to clinical examination and screening blood tests, including full blood count (FBC), urea and electrolytes (U&E), and liver functions tests (LFT) - see exclusion criteria for further details

Exclusion Criteria:

* Use of any additional investigational medications or products within 28 days of screening (including prior to screening)
* Use of intra-muscular/intra-articular or oral corticosteroids within 28 days prior to screening
* Use (including use as required) of more than one NSAID, change in NSAID or change in dose of NSAID within 28 days of the baseline visit.
* Live vaccine within <28 days prior to screening
* Pregnant/lactating women or planning pregnancy within 24 weeks of last protocol treatment
* Planned surgery within the study period (requiring omission of study medication > 28 days
* The presence of other comorbidities, which the physician deems as significant to interfere with evaluation (musculoskeletal condition such as osteoarthritis & fibromyalgia)
* Diagnosis of another inflammatory arthritis or connective tissue disease (e.g. psoriatic arthritis or Ankylosing spondylitis, primary Sjogren's syndrome, systemic sclerosis, systemic lupus erythematosus, polymyositis)
* Concomitant severe infection requiring intravenous therapy 4 weeks (28) days prior to screening
* Any contraindication to conventional DMARD's/anti-TNF therapy
* Patients with abnormal liver function at the time of screening or abnormal blood tests as shown by:

  * Aminotransferase (AST) / alanine aminotransferase (ALT) > 3x upper limit of normal (ULN) OR Bilirubin > 50µmol/L
  * Serum Creatinine > 175 umol/L
  * eGFR below 30ml/L/min/1.73m2
  * neutrophils < 2000 x 106/L
  * Platelets < 125 x 109/L
  * Haemoglobin < 90 g/L for males and < 85 g/L for females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission at 24 weeks (Arms A vs B) | 24 weeks
  The difference in the proportions of patients in clinical remission (DAS28ESR ≤2.6) at 24 weeks of first-line methotrexate with T2T care between those with normal (Arm A) vs. abnormal (Arm B) naïve CD4+ T-cell frequencies

SECONDARY OUTCOMES:
Clinical Remission at 12 weeks (Arms A vs B) | 12 weeks
  The difference in the proportions of patients in clinical remission (DAS28ESR ≤2.6) after 12 weeks of first-line methotrexate with T2T care between those with normal (Arm A) vs. abnormal (Arm B) naïve CD4+ T-cell frequencies
Clinical Remission at 12 and 24 weeks (Arms B vs C) | 12 and 24 weeks
  The difference in the proportions of patients in clinical remission (DAS28ESR ≤2.6) at 12 weeks and 24 weeks for patients with abnormal baseline naïve CD4+ T-cell frequencies receiving methotrexate with T2T care (Arm B) vs. etanercept + methotrexate (Arm C)
Sustained Clinical Remission | 12 and 24 weeks
  The difference in the proportions of patients achieving sustained clinical remission (DAS28ESR ≤2.6 at both 12 and 24 weeks) (Arm A vs. Arm B and Arm B vs. Arm C)
Patient Reported Outcomes at 12 and 24 weeks (Arm A vs B) | 12 and 24 weeks
  The differences in the medians of patient-reported outcome measures (EMS, VAS scales, HAQ-DI) after 12 weeks & 24 weeks of first-line methotrexate with T2T care between those with normal (Arm A) vs. abnormal (Arm B) naïve CD4+ T-cell frequencies
Patient Reported Outcomes at 12 and 24 weeks (Arm B vs C) | 12 and 24 weeks
  The differences in the medians of patient-reported outcome measures (EMS, VAS scales, HAQ-DI) after 12 weeks & 24 weeks for patients with abnormal baseline naïve CD4+ T-cell frequencies receiving methotrexate with T2T care (Arm B) vs. etanercept + methotrexate (Arm C)
Imaging Remission at 24 weeks (Arm A vs B) | 24 weeks
  The difference in the proportions of patients in imaging remission (Total power doppler synovitis score=0) after 24 weeks of first-line methotrexate with T2T care between those with normal (Arm A) or abnormal (Arm B) naïve CD4+ T-cell frequencies
Imaging Remission at 24 weeks (Arm B vs C) | 24 weeks
  The difference in the proportions of patients in imaging remission (Total power doppler synovitis score = 0) at 24 weeks for patients with abnormal baseline naïve CD4+ T-cell frequencies receiving methotrexate with T2T care (Arm B) vs. etanercept + methotrexate (Arm C)
Immunological Remission | 24 weeks
  The difference in the proportion of patients with normal naïve CD4+ T-cells at 24 weeks for patients with abnormal baseline naïve CD4+ T-cells receiving methotrexate with T2T care (Arm B) vs. etanercept + methotrexate (Arm C)
Cumulative Steroid Use | 24 weeks
  The difference in the average (median) cumulative amount of intramuscular corticosteroid use at 24 weeks between study arms (Arm A vs. Arm B and Arm B vs. Arm C). This will include any administered at the 24 week visit.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Emery, Professor, Principal Investigator — Institute of Rheumatic & Musculoskeletal Medicine, Chapel Allerton Hospital
Locations (1):
- Institute of Rheumatic & Musculoskeletal Medicine, Chapel Allerton Hospital, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided